CLINICAL TRIAL: NCT03302962
Title: Factors Influencing Pediatric Asthma
Acronym: FIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Missouri Breaks Industries Research, Inc. (Other)
Collaborators: Sanford Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1U54MD008164-01 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Asthma in Children
Keywords: asthma; pediatric; american indian; children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Asthma Education (Experimental): One half (54) of the identified cases were randomized to receive the previously established "BREATHE" study educational program, emphasizing patient-centered, self management of asthma. Periodic follow-up through personal contact and surveillance of IHS RPMS or other medical provider records was conducted.
  Interventions: Behavioral: Intensive Asthma Education
- Routine Asthma Education Literature (No Intervention): The remaining 54 cases were randomized to the "control" arm and received written materials related to patient-centered asthma control.

INTERVENTIONS:
Behavioral: Intensive Asthma Education — One half (54) of the identified cases were randomized to receive the previously established "BREATHE" study educational program, emphasizing patient-centered, self management of asthma. Periodic follow-up through personal contact and surveillance of IHS RPMS or other medical provider records was conducted.
  Arms: Intensive Asthma Education

SUMMARY:
Asthma is a chronic lung disease with serious morbidity and potential mortality. Multiple physiologic, environmental and social conditions impact the prevalence and severity of asthma. Even when diagnosed, effective control can be impeded by improper use of medication, not understanding or being unable to avoid environmental triggers, lack of continuity in follow-up care, and lack of an asthma action plan. American Indians are especially at-risk for health problems related to asthma. American Indians have the highest asthma rate among single-race groups; 18.5% of American Indians are diagnosed with asthma, while only 11% are diagnosed with asthma in the general population but little is known about why this is true. Asthma is a prototypic example of the interaction of biologic, environmental and psychosocial influences on disease and this study investigated the possible improvement in asthma control from an intensive educational intervention.

DETAILED DESCRIPTION:
The primary aim of this study was to test the hypothesis that intensive patient education regarding self-directed, stepped care will result in reduced morbidity and medical care utilization, while increasing quality of life.

One half (54) of the identified cases will be randomized to receive the previously established "BREATHE" study educational program, emphasizing patient-centered, self management of asthma. Periodic follow-up through personal contact and surveillance of IHS RPMS or other medical provider records was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Cases must be "American Indian" (eligibile for care within the Indian Health Service); and at least 2 of the following 3 criteria:

  1. a diagnosis of asthma on at least 2 occasions by more than one provider during the past 2 years.
  2. refills of asthma treatment medications on at least 2 occasions during the past 2 years.
  3. Improvement of spirometry FEV1 of 20% with use of albuterol MDI or nebulizer.
* Controls meet the same demographic criteria as cases, but must also meet all of the following criteria.

  1. No diagnosis of asthma by any provider during the past 2 years.
  2. No prescriptions of any asthma meds during the past 2 years.
  3. FEV1 on spirometry greater than 80% of predicted value Exclusion Criteria:

Exclusion Criteria:

1. Birthweight less than 2500 grams
2. Neonatal ventilator treatment
3. Hospitalization at birth greater than 15 days.
4. Congenital heart anomaly requiring surgery
5. Diagnosis of cystic fibrosis
6. Congenital lung, diaphragm, chest wall, or airway anomaly
7. Diagnosis of pneumonia, pertussis, or tuberculosis within the past year
8. Congenital muscular disorder

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Chart Review of ED Visits | 3 years
  Emergency room visits for pulmonary complaints

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Breaks Industries Research Inc., Eagle Butte, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
This study was conducted by permission of the Cheyenne River Sioux Tribe and data sharing is allowed only with their permission. Any investigators wishing to access data from the study should contact Missouri Breaks Industries Research Inc for information on application procedures.